CLINICAL TRIAL: NCT02442063
Title: An Open-label, Multi-center, Non-randomized Phase Ib Study to Investigate Safety and Tolerability of Radium Ra 223 Dichloride (BAY88-8223) Administered in Combination With Paclitaxel in Cancer Subjects With Bone Lesions
Brief Title: Phase Ib Study of Radium Ra 223 Dichloride in Combination With Paclitaxel in Cancer Subjects With Bone Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 17110; 2015-000083-34 (EudraCT Number)
Record Dates: First submitted 2015-05-04; First posted 2015-05-13 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms; Bone Diseases
MeSH Terms: conditions — Neoplasms; Bone Diseases | interventions — radium Ra 223 dichloride; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radium Ra 223 dichloride (Experimental): Radium Ra 223 dichloride (Xofigo, BAY88-8223)
  Interventions: Drug: Radium Ra 223 dichloride (Xofigo, BAY88-8223); Drug: paclitaxel

INTERVENTIONS:
Drug: Radium Ra 223 dichloride (Xofigo, BAY88-8223) — 50 kBq/kg intravenous injection once every 4 weeks, will be administrated from cycle 2 up to 6 cycles
Drug: paclitaxel — 90 mg/m2 intravenous injection per week in a 3-week-on / 1-week-off regimen, will be administered as per local standard of care, starting in cycle 1

SUMMARY:
This phase Ib combination study is being conducted to assess the safety and tolerability of radium Ra 223 dichloride in combination with paclitaxel in cancer subjects with bone lesions with special focus on Grade 3/4 incidence of neutro- and/or thrombocytopenia and exploration of the mode of interaction (i.e. additive or synergistic interaction) between the selected chemotherapy and radium Ra 223 dichloride with regard to myelosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Subjects diagnosed with histologically or cytologically confirmed malignant solid tumors and at least two according bone lesions. A standard of practice bone scan for the documentation of at least 2 bone lesions can be used as long as it is within 3 months of planned start of treatment. If no bone scan within a 3 month window is available, then technetium 99m or NaF PET bone scan will be obtained at screening (within 28 days of planned start of study drug)
* Eligible to treatment with paclitaxel as single agent, following the assessment of the investigator. If treatment with paclitaxel has already been initiated before signing the informed consent, patients will not be eligible.
* For women: documentation of menopausal status: pre menopausal or post menopausal subjects. Post menopausal status is defined either by: one year or more of amenorrhea in the absence of other biological or physiological causes, or surgical menopause with bilateral oophorectomy.
* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the informed consent form and for 6 months after the last radium Ra 223 dichloride administration. These procedures should be documented in source documents, the investigator or a designated associate is requested to advise the subject on how to achieve birth control.
* Women of childbearing potential must have a serum pregnancy test performed within 7 days before start of study treatment, and a negative result must be documented before start of study treatment
* Life expectancy of at least 16 weeks
* Adequate bone marrow function assessed within 7 days of starting the study treatment, judged by the following laboratory values:

  * Platelet count ≥ 100.000/cubic millimeters (mm3), within 7 days of starting the study treatment AND
  * Hemoglobin (HB) ≥ 9.0g/dl, within 7 days of starting the study treatment AND
  * Absolute neutrophil count (ANC) ≥ 1500/mm3 within 7 days of starting the study treatment
* Adequate liver function assessed within 7 days of starting the study treatment, judged by the following laboratory values:

  * Total bilirubin ≤ 1.5 x the upper limit of normal range (ULN) (except for subjects with documented Gilbert's disease) AND
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤5 x ULN for subjects whose cancer involves their liver including liver metastasis) within 7 days of starting the study treatment AND
  * Albumin > 30 g/L within 7 days of starting the study treatment
* International normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation. Patients being treated with anticoagulant, e.g. heparin, will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists and INR of the patient is < 3. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care If patients are on newer generation therapeutic blood thinning agents without the requirement of monitoring (e.g. Xarelto, Dabigatran), patients are eligible and management (e.g. discontinuation of the anticoagulant) will be handled by good medical practice standards under direction of the investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Estimated creatinine clearance (CLCr) ≥ 30 mL/min as calculated using the Cockcroft-Gault equation

Exclusion Criteria:

* History of other malignancy which could affect compliance with the protocol or interpretation of results.
* Received systemic therapy with radionuclides (e.g., strontium 89, samarium 153, rhenium 186, rhenium 188 or radium 223), including radium Ra 223 dichloride, for the treatment of bone metastases
* Previous (within 4 weeks prior to first treatment within this study) or concomitant participation in another clinical study with investigational medicinal product(s)
* Imminent or established spinal cord compression based on clinical findings and/or MRI.
* Active brain metastases or meningeal tumors if the subject is < 2 months from definitive therapy, has evidence of tumor growth on an imaging study within 4 weeks prior to study entry and is on dexamethasone and not clinically stable with respect to the tumor at the time of study entry.
* Prior hemibody external radiotherapy
* Bone fracture in weight bearing bones without acceptable orthopedic stabilization within 4 weeks prior to start of treatment
* Confirmed Paget's disease of the bone
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks) or pulmonary embolism within 6 months before the start of study medication or deep vein thrombosis within 3 months before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than 1 month before the start of study medication)
* Subjects with evidence or history of bleeding diathesis; any hemorrhage or bleeding event CTCAE Grade ≥ 3 or higher within 4 weeks of start of investigational treatment
* History of Bone marrow dysplasia
* Pregnancy and lactation (breast feeding)
* Evidence of peripheral neuropathy > grade 1
* Blood transfusion or use of erythropoietin within 6 weeks prior to start of study treatment (chemotherapy). Platelet transfusions are not allowed within 3 weeks prior to start of study treatment (chemotherapy). Use of biologic response modifies, such as granulocyte macrophage-colony-stimulating factor (GM-CSF or granulocyte-colony-stimulating factor (G-CSF), within 6 weeks prior to start of study treatment (chemotherapy).
* Intake of clozapine within 4 weeks before start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The percentage of participants with thrombocytopenia during cycle 1 (paclitaxel alone), 2 and 3 (combination treatment) | Approximately 12 weeks
The percentage of participants with neutropenia during cycle 1 (paclitaxel alone), 2 and 3 (combination treatment) | Approximately 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- HUS, Finland
- Israel (2):
  - Haifa
  - Tel Aviv
- United Kingdom (2):
  - Sutton, Surrey
  - Sheffield